CLINICAL TRIAL: NCT04577768
Title: The Effect of Transcranial Direct Current Stimulation Intensity on Motor Performance in Healthy Adults
Brief Title: The Effect of Transcranial Direct Current Stimulation on Motor Performance in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ariel University (Other)
Collaborators: Tel Aviv University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AU-HEA-SFT-20190326
Record Dates: First submitted 2020-09-23; First posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-09

CONDITIONS: Healthy
Keywords: transcranial direct current stimulation; motor performance

STUDY DESIGN:
Intervention Model Description: randomized controlled trial (RCT)
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HD-tDCS 2 mA (Experimental): Single session of 20-min HD-tDCS to the right primary motor cortex with an intensity of 2 mA. The session lasted approximately one hour. The participants returned after 24 hours to perform a retention test.
  Interventions: Device: HD-tDCS 2 mA
- HD-tDCS 1.5 mA (Experimental): Single session of 20-min HD-tDCS to the right primary motor cortex with an intensity of 1.5 mA. The session lasted approximately one hour. The participants returned after 24 hours to perform a retention test.
  Interventions: Device: HD-tDCS 1.5 mA
- Control (Sham Comparator): Single session of 20-min of sham HD-tDCS. The session lasted approximately one hour. The participants returned after 24 hours to perform a retention test.
  Interventions: Device: HD-tDCS sham

INTERVENTIONS:
Device: HD-tDCS 2 mA — anodal high definition transcranial direct current stimulation of the right primary motor cortex with an intensity of 2 mA
  Arms: HD-tDCS 2 mA
Device: HD-tDCS 1.5 mA — anodal high definition transcranial direct current stimulation of the right primary motor cortex with an intensity of 1.5 mA
  Arms: HD-tDCS 1.5 mA
Device: HD-tDCS sham — sham stimulation of the right primary motor cortex
  Arms: Control

SUMMARY:
to investigate the effect of stimulation intensity on motor performance in healthy adults.

DETAILED DESCRIPTION:
60 healthy subjects were randomly allocated to one of three groups: (a) 20-min of High-Definition transcranial direct current stimulation (HD-tDCS) with an intensity of 2 mA (HD-tDCS 2 mA); (2) 20-min of HD-tDCS with an intensity of 1.5 mA (HD-tDCS 1.5 mA); and (3) 20-min of sham HD-tDCS (HD-tDCS sham). The stimulation was administered noninvasively using an M x N 9-channel high definition transcranial electrical current stimulator from Soterix Medical (New York, NY). The anodal stimulation targeted the right Brodmann area 4 (primary motor cortex) based on HD-Targets brain modelling software (Soterix Medical, New York, NY).

Tests: The non-dominant left arm was tested. The subjects performed a sequential point-to-point movement task on the graphics tablet. Initially, the participants were required to perform 3 sequences without errors to familiarize themselves with the setup, the task and the sequence. Then, they performed the pre-test which consisted of two blocks of 6 sequences, i.e. 12 sequences, with a 30 s break between blocks. Two min after starting the appropriate stimulation, they performed 2 blocks of 6 sequences (identical to the pre-test). After finishing the tDCS stimulation, the participants performed a post-test, which was also identical to the pre-test. The participants returned after 24 hours to perform a retention test, which was equivalent to the pre- and post-tests. Two outcome measures were used: movement time (s) and the reaction time (s) of the reaching movements.

ELIGIBILITY:
Inclusion Criteria:

* aged between 20 and 35
* right-hand dominant
* healthy according to self report

Exclusion Criteria:

* taking psychiatric medications
* a history of drug abuse or dependence
* psychiatric or neurological disorder
* a history of seizures
* metal implants in their head
* musculoskeletal deficits interfering with task performance (proper reaching performance in sitting)

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-07-11 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
Change in movement time (s) from baseline to intervention | Baseline (immediately before stimulation), two minutes after starting the stimulation
  Time from movement onset (first time the tangential velocity was greater than 5% of the peak tangential velocity) until the end of the movement (the last time the tangential velocity was greater than 5% of the peak tangential velocity). Improved motor performance was indicated by a shorter movement time.
Change in movement time (s) from baseline to posttest | Baseline (immediately before stimulation), immediately post stimulation
  Time from movement onset (first time the tangential velocity was greater than 5% of the peak tangential velocity) until the end of the movement (the last time the tangential velocity was greater than 5% of the peak tangential velocity). Improved motor performance was indicated by a shorter movement time.
Change in movement time (s) from baseline to retention test | Baseline (immediately before stimulation), 24 hours following the stimulation
  Time from movement onset (first time the tangential velocity was greater than 5% of the peak tangential velocity) until the end of the movement (the last time the tangential velocity was greater than 5% of the peak tangential velocity). Improved motor performance was indicated by a shorter movement time.
Change in movement time (s) from intervention to posttest | Two minutes after starting the stimulation, immediately post stimulation
  Time from movement onset (first time the tangential velocity was greater than 5% of the peak tangential velocity) until the end of the movement (the last time the tangential velocity was greater than 5% of the peak tangential velocity). Improved motor performance was indicated by a shorter movement time.
Change in movement time (s) from intervention to retention test | Two minutes after starting the stimulation, 24 hours following the stimulation
  Time from movement onset (first time the tangential velocity was greater than 5% of the peak tangential velocity) until the end of the movement (the last time the tangential velocity was greater than 5% of the peak tangential velocity). Improved motor performance was indicated by a shorter movement time.
Change in movement time (s) from posttest to retention test | immediately post stimulation, 24 hours following the stimulation
  Time from movement onset (first time the tangential velocity was greater than 5% of the peak tangential velocity) until the end of the movement (the last time the tangential velocity was greater than 5% of the peak tangential velocity). Improved motor performance was indicated by a shorter movement time.
Change in reaction time (s) from baseline to intervention | Baseline (immediately before stimulation), two minutes after starting the stimulation
  Time between when the target appeared in green (changed color from white to green), and movement onset. Improved motor performance was indicated by a shorter reaction time.
Change in reaction time (s) from baseline to posttest | Baseline (immediately before stimulation), immediately post stimulation
  Time between when the target appeared in green (changed color from white to green), and movement onset. Improved motor performance was indicated by a shorter reaction time.
Change in reaction time (s) from baseline to retention test | Baseline (immediately before stimulation), 24 hours following the stimulation
  Time between when the target appeared in green (changed color from white to green), and movement onset. Improved motor performance was indicated by a shorter reaction time.
Change in reaction time (s) from intervention to posttest | Two minutes after starting the stimulation, immediately post stimulation
  Time between when the target appeared in green (changed color from white to green), and movement onset. Improved motor performance was indicated by a shorter reaction time.
Change in reaction time (s) from intervention to retention test | Two minutes after starting the stimulation, 24 hours following the stimulation
  Time between when the target appeared in green (changed color from white to green), and movement onset. Improved motor performance was indicated by a shorter reaction time.
Change in reaction time (s) from posttest to retention test | immediately post stimulation, 24 hours following the stimulation
  Time between when the target appeared in green (changed color from white to green), and movement onset. Improved motor performance was indicated by a shorter reaction time.

CONTACTS AND LOCATIONS:
Overall Officials: Silvi Frenkel-Toledo, Principal Investigator — Ariel University
Locations (1):
- Ariel University, Ariel, Israel

IPD SHARING:
Plan to Share IPD: No
The datasets (Study Protocol, Statistical Analysis Plan, Informed Consent Form, Analytic Code generated during and/or analyzed during the current study) are available from the corresponding author on reasonable request.

REFERENCES:
- [Derived] Lerner O, Friedman J, Frenkel-Toledo S. The effect of high-definition transcranial direct current stimulation intensity on motor performance in healthy adults: a randomized controlled trial. J Neuroeng Rehabil. 2021 Jun 26;18(1):103. doi: 10.1186/s12984-021-00899-z. PMID 34174914